CLINICAL TRIAL: NCT05374590
Title: A Long-term, Single-Arm, Open-label, Multicenter Trial to Evaluate Safety of Efgartigimod Administered Intravenously and Efgartigimod PH20 Administered Subcutaneously in Children With Generalized Myasthenia Gravis
Brief Title: Evaluating Long-term Safety of Efgartigimod Administered Intravenously and Efgartigimod PH20 Administered Subcutaneously in Children With Generalized Myasthenia Gravis
Acronym: ADAPT Jr +
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2008; 2023-507379-23-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-01; First posted 2022-05-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis; gMG
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Efgartigimod or Efgartigimod PH20 SC (Experimental): Patients receiving Efgartigimod IV treatment or Efgartigimod PH 20 SC treatment
  Interventions: Biological: Efgartigimod IV or Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod IV or Efgartigimod PH20 SC — Intravenous infusion of Efgartigimod or Subcutaneous injection of Efgartigimod PH20 SC

SUMMARY:
The purpose of this trial is to evaluate the long-term safety of efgartigimod IV and efgartigimod PH20 SC administered to participants with gMG in the antecedent studies, ARGX-113-2006 and ARGX-113-2207, respectively.

Participants will receive efgartigimod IV or efgartigimod PH20 SC, using the dose administered in the antecedent studies. Participants who have not reached the age of 18 can remain in the study until efgartigimod becomes commercially available in the respective country or available through another continued access program for gMG. Participants who have reached the age of 18 can remain in the study for a maximum of 2 years, until efgartigimod becomes commercially available in the respective country or available through another continued access program for gMG, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* The participant completed ARGX-113-2006, defined as:

  1. The participant reached End of Trial in trial ARGX-113-2006 or End of Study in ARGX-113-2207 and agreed to participate in the ARGX-113-2008 trial.
  2. The participant qualifies for retreatment in trial ARGX-113-2006, but cannot complete a Treatment Period (TP) and the required Intertreatment Period (IP) visits within the ARGX-113-2006 trial's timeframe.
* Either the participant or the participant's legally authorized representative can understand the requirements of the trial and provide written informed consent/assent, and willingness and ability to comply with the trial protocol procedures.
* Contraceptive use for sexually active participants should be consistent with local regulations for those participating in clinical studies.

Exclusion Criteria:

* Female adolescents of childbearing potential (FAOCBP): Pregnancy or lactation, or the participant intends to become pregnant during their participation in the study.
* Discontinued early from ARGX-113-2006 or ARGX-113-2207 treatment.
* Clinically significant uncontrolled chronic bacterial, viral, or fungal infection at study entry not sufficiently resolved in the investigator's opinion or known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of gMG or put the participant at undue risk.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs and AESIs | Up to 4 years
  AE : adverse event; SAE : serious adverse event; AESI : adverse event of special interest

SECONDARY OUTCOMES:
Incidence of ADAs against efgartigimod | Up to 4 years
  ADA : anti-drug antibody
Incidence of antibodies against rHuPH20 | Up to 4 years
  rHuPH20: recombinant human hyaluronidase PH20

CONTACTS AND LOCATIONS:
Locations (16):
- United States (3):
  - Ann and Robert H Lurie Children's Hospital of Chicago - Main Hospital, Chicago, Illinois
  - Atrium Health Neurology Specialty Care, Charlotte, North Carolina
  - University of Virginia (UVA) Health - Developmental Pediatrics Clinic, Charlottesville, Virginia
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
- Childrens Hospital of Eastern Ontario, Ottawa, Canada
- AP-HM- Hôpital de La Timone, Marseille, France
- Universitätsklinikum Essen, Essen, Germany
- Hadassah Medical Center- Ein Kerem, Jerusalem, Israel
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne w Gdansku, Gdansk
  - Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Centralny Szpital Kliniczny - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
- Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Spain
- United Kingdom (2):
  - Great Ormand Street Hospital for Children NHS Foundation Trust - Great Ormond Street Hospital - Pediatric Neurology, London
  - Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital Children's Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided